CLINICAL TRIAL: NCT01717976
Title: Discharge Information & Support for Patients Receiving Outpatient Care in the ED
Brief Title: Discharge Information and Support for Patients Receiving Outpatient Care in the Emergency Department
Acronym: DISPO ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IIR 12-052
Record Dates: First submitted 2012-10-26; First posted 2012-10-31 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-06

CONDITIONS: Multimorbidity
Keywords: emergency department use; Veterans

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): primary care based nurse telephone support
  Interventions: Behavioral: DISPO ED
- Control (No Intervention): usual care

INTERVENTIONS:
Behavioral: DISPO ED — primary care based nurse telephone support
  Arms: Intervention

SUMMARY:
The Veterans' Health Administration (VHA) is committed to improving primary care through the implementation of Patient Aligned Care Teams (PACTs). Improving access to services and care coordination are among the primary goals of PACTs; however, there remain many unanswered questions about how best to use the limited time of PACT team members, such as nurse care managers, to accomplish this. This study will evaluate the effectiveness of a nurse-led telephone support program for Veterans who have been treated recently in the emergency department (ED) and are at high risk for repeat visits. The program's goals are to reduce the need for future ED use and improve satisfaction among Veterans by providing information and support related to the ED visit, enhancing chronic disease management and educating Veterans and family members about PACT and other VA and community services. If proven effective, this program could improve health and healthcare for a large, vulnerable group of Veterans and be cost saving for VHA.

DETAILED DESCRIPTION:
Anticipated Impacts on Veteran's Healthcare More than 1 million Veterans receive care in Emergency Departments (EDs) in VA Medical Centers (VAMCs) annually. ED visits that do not result in hospital admission, commonly referred to as treat and release visits, account for 80% of all VAMC ED encounters. Nearly 1 in 5 Veterans treated and released from a VAMC ED receive additional unscheduled care in the ED or hospital within 30 days, a rate that is higher than non-VA settings. A large number of Veterans and the VA system would benefit from the development of interventions that reduce subsequent ED use in this vulnerable population.

Project Background Failing to address unmet needs and difficulty navigating the health system are two primary forces driving repeat ED use. Unmet needs after an ED visit range from poorly controlled chronic diseases to incomplete understanding of new medications or follow-up instructions. Perceived barriers to access to primary care and other services are also cited as factors that lead Veterans back to the ED for ambulatory care. In a nationally representative sample of 15,263 Veterans with repeat ED visits, the investigators found that 71.7% did not see another VA outpatient provider between their original and return trip to the ED, Improving access to services and care coordination are among the primary goals of the Veterans' Health Administration's (VHA) ongoing reorganization of primary care. Patient Aligned Care Teams (PACTs) are being created in VAMCs across the country; however, there has been little focus on the interface between PACT and the ED. A key role for nurses within PACT will be telephone management of high risk populations, and Veterans treated and released from the ED represent one such high-risk group. However, no studies have examined both the Veteran and system-level impact of using nurse care managers to support Veterans after an ED visit.

Project Objectives

The overall goal of this study is to examine the impact of a primary care-based nurse telephone support program for Veterans treated and released from the ED who are at high risk for repeat visits. The investigators will test the following hypotheses:

H1: Veterans who participate in a primary care-based nurse telephone support program after an ED visit will have fewer ED visits in the subsequent 30 days compared to usual care;

H2: Veterans who participate in a primary care- based nurse telephone support program after an ED visit will have higher satisfaction compared to usual care;

H3: Veterans who participate in a primary care-based nurse telephone support program will have lower VA costs for ED and hospital care in the 180 days following an ED visit, compared to usual care.

Project Methods The proposed study is a two group randomized, controlled trial to evaluate a structured nurse telephone support program for Veterans treated and released from the ED who are at high risk for repeat visits. After informed consent is obtained, Veterans will be randomized to nurse telephone support [DISPO ED] or usual care. DISPO ED will consist of 2 calls from a study nurse (simulating the role of a PACT RN Care Manager) within 7 days of the index ED visit, with an option for a 3rd call within 14 days. The primary outcome is a dichotomous outcome defined as any ED use within 30 days or not. Secondary outcomes are patient satisfaction with VA health care at 30 and 180 days, and total VA costs within 180 days.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, patients must meet all of the following:

* Treated and released from the Durham VA ED;
* Receive primary care from a Durham VAMC affiliated primary care clinic (at least one visit in a primary care clinic affiliated with the Durham VAMC within the previous 12 months);
* At least one VAMC ED visit or hospital admission within the 6 months preceding the index visit;
* Diagnosed with 2 or more chronic health conditions; and
* Valid telephone number in the medical record; in the investigators' pilot studies, 98.7% of Veterans had a valid phone number in the medical record.

Exclusion Criteria:

Patients will be excluded if they meet any of the following:

* Reside in a nursing home (or other institutional setting);
* Unable to communicate on the telephone, and no proxy available;
* Lacks decision-making capacity, and no proxy available; or
* Returned to ED within 24 hours of discharge from initial visit.
* Have a current Category 1 high-risk suicide flag on their CPRS medical record; or Visit the PEC (Psychiatric Emergency Clinic) within 24 hours of discharge from initial ED visit.
* Enrolled in a study that prohibits cross-enrollment in other studies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2013-12; Primary Completion 2016-03 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan N. Hastings, MD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hastings SN, Betts E, Schmader KE, Weinberger M, Van Houtven CH, Hendrix CC, Coffman CJ, Stechuchak KM, Weiner M, Morris K, Kessler C, Oddone EZ. Discharge information and support for veterans Receiving Outpatient Care in the Emergency Department: study design and methods. Contemp Clin Trials. 2014 Nov;39(2):342-50. doi: 10.1016/j.cct.2014.10.008. Epub 2014 Nov 3. PMID 25445314
- [Derived] Seidenfeld J, Ramos K, Bruening RA, Sperber NR, Stechuchak KM, Hastings SN. Patient experiences of a care transition intervention for Veterans to reduce emergency department visits. Acad Emerg Med. 2023 Apr;30(4):388-397. doi: 10.1111/acem.14661. Epub 2023 Jan 30. PMID 36630213
- [Derived] Ramos K, Shepherd-Banigan ME, Stechuchak KM, Coffman C, Oddone EZ, Van Houtven C, Hendrix CC, Mahanna EP, Hastings SN. Psychological distress among medically complex veterans with a recent emergency department visit. Psychol Serv. 2022 May;19(2):353-359. doi: 10.1037/ser0000437. Epub 2021 Apr 1. PMID 33793285
- [Derived] Hastings SN, Stechuchak KM, Coffman CJ, Mahanna EP, Weinberger M, Van Houtven CH, Schmader KE, Hendrix CC, Kessler C, Hughes JM, Ramos K, Wieland GD, Weiner M, Robinson K, Oddone E. Discharge Information and Support for Patients Discharged from the Emergency Department: Results from a Randomized Controlled Trial. J Gen Intern Med. 2020 Jan;35(1):79-86. doi: 10.1007/s11606-019-05319-6. Epub 2019 Sep 5. PMID 31489559

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 514 participants were randomized and assigned to either DISPO ED or usual care. One participant (UC arm) was found to be ineligible post-randomization and thus not included in analyses.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 257 | 257
Completed | 257 | 256
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 257 | 256 | 513
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (12.7) | 59.4 (11.5) | 59.1 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 54 | 114
  Male | 197 | 202 | 399

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Repeat ED Use
Description: Number of Participants Experiencing Repeat ED Use
Time Frame: 30 days
Population: 0 out of the 257 participants in the DISPO intervention group and 1 of the 256 participants in the Usual Care group were deceased at 30 days and not included in the primary outcome analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 257 | 255
Participants | 64 | 59

2. Secondary Outcome: Number of Participants Satisfied With Health Care
Description: Satisfaction with health care determined by 9 or 10 on the CAHPS
Time Frame: Baseline
Population: 0 out of 257 in intervention group and 2 out of 256 participants in the usual care group had missing data at baseline for satisfaction due to non-response.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 257 | 254
Participants | 110 | 117

3. Secondary Outcome: Number of Participants Satisfied With Health Care
Description: Satisfaction with health care determined by 9 or 10 on the CAHPS
Time Frame: 30 days
Population: 24 out of 257 in intervention group and 38 out of 256 participants in the usual care group had missing data at the 30 day interview for satisfaction due to missing the 30-day interview or non-response to the satisfaction question at the 30 day interview.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 233 | 218
Participants | 117 | 109

4. Secondary Outcome: Number of Participants Satisfied With Health Care
Description: Satisfaction with health care determined by 9 or 10 on the CAHPS
Time Frame: 180 days
Population: 26 out of 257 in intervention group and 33 out of 256 participants in the usual care group had missing data at the 180 day interview for satisfaction due to missing the 180-day interview or non-response to the satisfaction question at the 180 day interview.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 231 | 223
Participants | 115 | 106

5. Secondary Outcome: Total Costs to the VHA
Description: Assessment of VA and VA purchased care costs in 2016 dollars within 180 days from emergency department visit
Time Frame: 180 days
Population: 0 out of 257 participants in the DISPO intervention group and 1 of 256 in the usual care group were deceased at 30 days and not included in the cost analysis.
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | Intervention | Control
Number analyzed (Participants) | 257 | 255
US Dollars | 38273.16 (57836.31) | 31696.00 (46294.63)

ADVERSE EVENTS:
Description: Adverse events were collected without regard to the specific Adverse Event Term.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 2/257 | 3/256
Serious Adverse Events (participants affected / at risk) | 18/257 | 21/256
Other Adverse Events (participants affected / at risk) | 0/257 | 0/256
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=257) | Control (N=256)
Hospitalizations (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hospitalizations (Cardiac disorders) | 5 (8) | 6 (6)
Hospitalizations (Gastrointestinal disorders) | 2 (2) | 2 (2)
Hospitalizations (General disorders) | 0 (0) | 2 (2)
Hospitalizations (Infections and infestations) | 0 (0) | 2 (2)
Hospitalizations (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Hospitalizations (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hospitalizations (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hospitalizations (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hospitalizations (Psychiatric disorders) | 1 (1) | 3 (3)
Hospitalizations (Renal and urinary disorders) | 0 (0) | 1 (1)
Hospitalizations (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hospitalizations (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hospitalizations (Surgical and medical procedures) | 1 (1) | 4 (4)
Hospitalizations (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes